CLINICAL TRIAL: NCT04377386
Title: Efficacy of Oral Vitamin D Supplementation in Reducing Body Mass Index and Lipid Profile in Adolescents and Young Adults in Colombia: a Pilot Clinical Trial Protocol Nested in the SIMBA Cohort
Brief Title: Efficacy of Oral Vitamin D Supplementation in Adolescents and Young Adults.
Acronym: SIMBAIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Universidad Industrial de Santander (Other); Farma de Colombia SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECA-SIMBA-III-2020; 656680763838 (Other Grant/Funding Number: COLCIENCIAS); 2020-03-71 (Other Grant/Funding Number: Universidad Industrial de Santander UIS); 133-052018 (Other Grant/Funding Number: Fundación Cardiovascular de Colombia)
Record Dates: First submitted 2020-04-07; First posted 2020-05-06 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity; Overweight Adolescents; Vitamin D Deficiency
Keywords: Vitamin D; Obesity; Weight loss; Body composition; Cholesterol; Triglycerides
MeSH Terms: conditions — Overweight; Obesity; Vitamin D Deficiency; Weight Loss | interventions — Cholecalciferol; Dietary Supplements; Vitamin D

STUDY DESIGN:
Intervention Model Description: Pilot study of a two-arm, triple-blind, parallel randomized controlled clinical trial, in 150 adolescents and young adults in the city of Bucaramanga-Colombia. All participants will be given 105 doses of VD. The 75 participants assigned to the intervention group will take one 1000 IU VD capsule daily for 15 weeks. On the other hand, the 75 participants in the control group will take 1 capsule of VD of 200 IU for the same time. The participants in both the intervention and the control group must record in a calendar the time of the daily intake of the supplement during the 15 weeks.
  The main outcomes are: serum levels of 25 (OH) D, body mass index and lipid profile; Secondary measures complement the previous ones (skin folds, waist-to-hip ratio). Other variables will be analyzed such as: assessment of dietary intake, physical activity, sun exposure, cigarette and tobacco consumption and adherence to supplementation with DV.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment of treatment in real time will be made with the support of a computer program. The procedure will take place by means of a single assignment sequence that determines the assignment code for each participant's treatment. This process allows all participants in the study to be assigned to any of the treatment groups.
  Supplements will be packaged in individual packages with the total number of doses per participant (105 doses). The coding of the packages will be in charge of the laboratory in charge of providing the supplements, which in turn will send to the designated person at the data center by institutional e-mail, a document with the list of codes and the dose of the supplement.
  The 1000 IU and 200 IU doses of VD will be provided in white containers and will be identical in terms of physical and organoleptic characteristics, to ensure that both participants and investigators are blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: 1000 IU DV (Experimental): The 75 participants assigned to the intervention group will take 1 DV capsule of 1000 IU daily for 15 weeks.
  Interventions: Dietary Supplement: 1000 IU D vitamin
- Control group: 200 IU DV (Placebo Comparator): The 75 participants of the control group will take 1 DV capsule of 200 IU daily for 15 weeks, this dose being the minimum recommended for children. The above, considering that it is ethical for the control group to receive a minimum dose of supplementation.
  Interventions: Dietary Supplement: 200 IU D vitamin

INTERVENTIONS:
Dietary Supplement: 1000 IU D vitamin — Participants in the intervention group will receive 105 DV doses of 1000 IU. The supplementation will be given by the Farma de Colombia laboratory, known commercially as Farma D, whose presentation is in soft gelatin capsules. It is recommended to take one dose per day at the same time and participants should record the daily intake time of the supplement for 15 weeks on a calendar.
  Other Names: Supplementation with 1000 IU vitamin D; Farma D 1000 IU
  Arms: Intervention group: 1000 IU DV
Dietary Supplement: 200 IU D vitamin — Participants in the control group will receive 105 DV doses of 200 IU. The supplementation will be given by the same laboratory; it will have the same characteristics and recommendations for the intake as for the intervention group.
  Other Names: Supplementation with 200 IU vitamin D; Farma D 200 IU
  Arms: Control group: 200 IU DV

SUMMARY:
This study assesses whether oral supplementation with vitamin D contributes to the reduction of body mass index and lipid profile in adolescents and young adults. The intervention group will receive 1000 IU of vitamin D (DV) and the control group 200 IU of DV.

DETAILED DESCRIPTION:
Sample size: the simple size was calculated considering the following parameters: an expected difference in the study outcomes (overweight, obesity, and alteration of the lipid profile) of 20% between the intervention group and the control group; a power of 90%, an alfa of 5%, an intervention group/control group ratio of 1:1, and a 20% adjustment for losses to follow-up, resulting in a sample of 270 participants (n=135 intervention and n=135 control group). The OpenEpi software was used for the calculation. Since this is a pilot study and considering the feasibility, the research team decided on a sample size of 150 participants (n=75 intervention group and n=75 control group).

Randomization and blinding: the randomization process will take place in two stages. An engineer from the data central will conduct the randomization of the list of the 217 potentially eligible participants by means of a computer program with random numbers and it will select 150 individuals to participate in the study. Subsequently, a nurse will make phone calls to schedule appointments and formalize the participation in the study, the signature of the informed consent, and the taking of baseline measures. Once these stages are concluded, the assignment of treatment in real time will be made with the support of a computer program. The procedure will take place by means of a single assignment sequence that determines the assignment code for each participant's treatment.

Supplements will be packaged in individual packages with the total number of doses per participant (105 doses). The coding of the packages will be in charge of the laboratory in charge of providing the supplements, which in turn will send to the designated person at the data center by institutional e-mail, a document with the list of codes and the dose of the supplement. The 1000 IU and 200 IU doses of VD will be provided in white containers and will be identical in terms of physical and organoleptic characteristics, to ensure that both participants and investigators are blinded to the treatment. To maximize adherence to the intervention, participants will be required to cross out daily supplementation on a calendar with the study period, which participants should return at the end of the study.

The results of the assignment will only be known by the systems engineer at the data center. In other words, this information "will not be visible" to the coordinating nurse, laboratory personnel in charge of processing biological samples, pediatrician, principal investigator of the study, or the epidemiologist in charge of quality control and data analysis. This will ensure the masking of the people in charge of measuring the outcomes, administering the intervention and analyzing the study data.

Recruitment: for recruitment, a study nurse in charge of enrollment will contact by phone the 217 successful participants of the third re-contact, explain the objective of the study and inquire about the interest to participate; if there is a positive response, inclusion and exclusion criteria will be verified. A list of eligible participants will be generated from the above process and sent to the person in charge of the randomization process.

After the randomization process, the study nurse will receive from the data center the list of the 150 participants selected, who will be invited to participate in the clinical trial. The nurse will call them on the pone for a face-to-face appointment where the details of the study will be informed, doubts will be clarified, and the informed consent form will be signed; a copy of the form will be given to the participant.

During that appointment, the collection of demographic and clinical data will take place, as well as a blood simple for further measurement of VD, lipid profile and glycaemia; The anthropometric nutritional, dietary and physical activity assessment will also be carried out. Once the baseline measurements are taken, the assignment to the intervention will be made in real time through software designed for the study.

Finally, the supplementation intervention will be explained in detail and the package corresponding to the participant's code will be delivered according to the process of assignment to the group (intervention/control), it will be clarified that the supplementation will last 15 weeks and then the second meeting will be scheduled to carry out again the measures taken at the beginning of the study. At the end, a third meeting will be scheduled for the delivery of results and recommendations.

Ethical considerations: the research will be carried out following the principles established in the Good Clinical Practice in Clinical Trials GPC/ICH. It is considered a minimum risk study according to resolution 008430 of October 4, 1993 of the Colombian Ministry of Health, since it includes the administration of a commonly used vitamin supplement with a wide therapeutic margin and for its administration the indications, doses and routes of administration established by the Institute for Drug and Food Surveillance (Invima, acronym in Spanish) are considered.

The vitamin supplement is supplied by the laboratory Farma de Colombia, commercially known as Farma D, whose presentation is in soft gelatin capsules and with registration number 2017 M-0012231-R1.

The processing of personal and clinical data and biological samples will be handled according to the Habeas Data Act (Act 1266 of 2008) of the government of Colombia.

The study was reviewed and endorsed by the Technical Scientific Committee (CTC) of Fundacion Cardiovascular de Colombia (FCV) according to minute N°133 of May 2018 and has the approval of the Research Ethics Committee (IEC) of the FCV according to minute N°480 of July 16, 2019.

The study nurse will explain the objectives, importance, risks, benefits of the research and the confidentiality of the data. Written informed consent will be given to study participants.

Statistical analysis : an analysis will be made by intention to treat. The description of the categorical variables will be made by means of absolute and relative values. Quantitative variables that present a normal distribution in Shapiro Wilk's test will be reported as mean and standard deviation, otherwise the median and interquartile range will be presented. The comparison of the basal characteristics of the study groups (intervention and control) will be done using the ratio comparison test (Chi-square or Fischer's exact test) and the Student's t-test or Mann-Whitney's U-test.

Quantitative outcome variables will be contrasted through paired t-tests or Wilcoxon tests for quantitative variables, methods of longitudinal data analysis will also be explored and for categorical ones the Mc Nemar test will be used. Statistical significance will be considered for all hypothesis tests when the p value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the SIMBA cohort.
* Age ≥ 18 years.
* Re-contact consent from previous studies.

Exclusion Criteria:

* Medical diagnosis of diabetes mellitus, clinically manifest endocrinopathies, acute or chronic infectious liver disease, and kidney disease.
* Adolescents or Young adults subject to treatment with steroids or hormones (except levothyroxine) up to one month before lab sample taking.
* Current supplementation with VD (any form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Change in body mass index between baseline and week 15 | Baseline and week 15
  Change in body mass index (BMI) will be made through of the measure of body weight will be in kilograms (kg) to one decimal place, and the size in meters (m) to two decimal places. From these measurements the body mass index will be obtained using the formula: BMI = Weight (kg) / size (m)2.
Change in lipid profile (Total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides) between baseline and week 15 | Baseline and week 15
  Serum is measured from the same blood samples drawn for vitamin D levels. The processing and analysis of the samples will be done respectively through enzymatic technique, selective liquid detergent, selective detergent accelerator and Glycerol Phosphate Oxidase.
Change in 25-hydroxyvitamin D [25(OH)D] levels between baseline and week 15 | baseline and week 15
  After a 10-12 hour fast, in peripheral venous blood 25-hydroxyvitamin D [25(OH)D] is quantified in serum by chemiluminescent microparticle immunoassay (CMIA).

SECONDARY OUTCOMES:
Change in waist - hip ratio between baseline and week 15 | Baseline and week 15
  Determines the intra-abdominal fat levels and is obtained by dividing the waist perimeter by the hip perimeter. The circumference of the waist shall be measured at the midpoint between the edge of the lower sack (10th rib) and the upper edge of the iliac crest, without adjusting or stopping touching the skin.
  For the measurement of the hip, the knees and the heels must be together; the most prominent part of the hip on both sides shall be located and the tape measure shall be passed following the same recommendations as for the circumference of the waist.
Change of percentage body fat (PBF) in skin folds between baseline and week 15 | Baseline and week 15
  These are taken for the indirect estimation by means of measuring the bicipital, tricipital, abdominal, and subscapular folds. These measurements will be taken using a Harpender® skinfold caliper. Percentage of body fat (%BF) calculated with the Siri equation for four skin folds (SF), like so: % BF SIRI = ((4.95 / D) - 4.5) x 100. Body density (D) is obtained using the linear regression equation proposed by Durnin and Womersley (C and D). D = C - M x log10 ∑ 4SF (bicipital, tricipital, abdominal, and subscapular).
Change in fasting blood glucose level between baseline and week 15 | Baseline and week 15
  After a 10-12 hour fast, blood glucose levels are measured in serum from the same blood samples drawn for vitamin D levels, using the hexokinase/G-6-PDH technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charoenngam N, Shirvani A, Holick MF. Vitamin D for skeletal and non-skeletal health: What we should know. J Clin Orthop Trauma. 2019 Nov-Dec;10(6):1082-1093. doi: 10.1016/j.jcot.2019.07.004. Epub 2019 Jul 13. PMID 31708633
- [Background] Al Mheid I, Quyyumi AA. Vitamin D and Cardiovascular Disease: Controversy Unresolved. J Am Coll Cardiol. 2017 Jul 4;70(1):89-100. doi: 10.1016/j.jacc.2017.05.031. PMID 28662812
- [Background] Gholami F, Moradi G, Zareei B, Rasouli MA, Nikkhoo B, Roshani D, Ghaderi E. The association between circulating 25-hydroxyvitamin D and cardiovascular diseases: a meta-analysis of prospective cohort studies. BMC Cardiovasc Disord. 2019 Nov 7;19(1):248. doi: 10.1186/s12872-019-1236-7. PMID 31699030
- [Background] Paschou SA, Kosmopoulos M, Nikas IP, Spartalis M, Kassi E, Goulis DG, Lambrinoudaki I, Siasos G. The Impact of Obesity on the Association between Vitamin D Deficiency and Cardiovascular Disease. Nutrients. 2019 Oct 14;11(10):2458. doi: 10.3390/nu11102458. PMID 31615154
- [Background] Alloubani A, Akhu-Zaheya L, Samara R, Abdulhafiz I, Saleh A, Altowijri A. Relationship between Vitamin D Deficiency, Diabetes, and Obesity. Diabetes Metab Syndr. 2019 Mar-Apr;13(2):1457-1461. doi: 10.1016/j.dsx.2019.02.021. Epub 2019 Feb 20. PMID 31336506
- [Background] Hossain MJ, Levinson A, George D, Canas J, Kumar S, Balagopal PB. Vitamin D Status and Cardiovascular Risk in Obesity: Effect of Physical Activity in Nonvitamin D Supplemented Adolescents. Metab Syndr Relat Disord. 2018 May;16(4):197-203. doi: 10.1089/met.2017.0171. Epub 2018 Mar 13. PMID 29649377
- [Background] Zakharova I, Klimov L, Kuryaninova V, Nikitina I, Malyavskaya S, Dolbnya S, Kasyanova A, Atanesyan R, Stoyan M, Todieva A, Kostrova G, Lebedev A. Vitamin D Insufficiency in Overweight and Obese Children and Adolescents. Front Endocrinol (Lausanne). 2019 Mar 1;10:103. doi: 10.3389/fendo.2019.00103. eCollection 2019. PMID 30881343
- [Background] Villa-Roel C, Buitrago A, Rodriguez DC, Cano DJ, Martinez MP, Camacho PA, Ruiz AJ, Duran AE. Prevalence of metabolic syndrome in scholars from Bucaramanga, Colombia: a population-based study. BMC Pediatr. 2009 Apr 21;9:28. doi: 10.1186/1471-2431-9-28. PMID 19383169
- [Background] Mueller NT, Pereira MA, Buitrago-Lopez A, Rodriguez DC, Duran AE, Ruiz AJ, Rueda-Clausen CF, Villa-Roel C. Adiposity indices in the prediction of insulin resistance in prepubertal Colombian children. Public Health Nutr. 2013 Feb;16(2):248-55. doi: 10.1017/S136898001200393X. Epub 2012 Aug 24. PMID 22916737
- [Background] Serrano N, Villa-Roel C, Gamboa-Delgado EM, Barrera JG, Quintero-Lesmes DC. Early evaluation of the metabolic syndrome in Bucaramanga, Colombia. Transl Pediatr. 2019 Dec;8(5):363-370. doi: 10.21037/tp.2019.04.04. PMID 31993348
- [Derived] Serrano NC, Rojas LZ, Gamboa-Delgado EM, Suarez DP, Salazar Acosta I, Romero SL, Forero M, Quintero-Lesmes DC. Efficacy of vitamin D supplementation in reducing body mass index and lipid profile in healthy young adults in Colombia: a pilot randomised controlled clinical trial. J Nutr Sci. 2023 Feb 22;12:e29. doi: 10.1017/jns.2022.108. eCollection 2023. PMID 36843975
- [Derived] Serrano NC, Romero SL, Suarez DP, Rojas LZ, Gamboa-Delgado EM, Forero M, Guio E, Quintero-Lesmes DC. Efficacy of oral Vitamin D supplementation in reducing body mass index and lipid profile in adolescents and young adults in Colombia: A pilot clinical trial protocol nested in the SIMBA cohort. Medicine (Baltimore). 2020 Aug 28;99(35):e21722. doi: 10.1097/MD.0000000000021722. PMID 32871891